CLINICAL TRIAL: NCT06337565
Title: Safety of IBD Drugs During Pregnancy and Breasfeeding: Mothers and Babies' Outcomes (DUMBO 2 Registry)
Brief Title: Safety of IBD Drugs During Pregnancy and Breasfeeding: Mothers and Babies' Outcomes
Status: Recruiting | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, María Chaparro Sánchez, Principal Investigator, gastroenterologist, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Other Study IDs: GIS-DUMBO 2-2024
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Drusgs for IBD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational study where pregnant women treated with non-anti-TNF agents or targeted small molecules approved for IBD treatment will be included. Although it is a multicentre, nationwide study, the number of patients to be included is expected to be relatively low (in DUMBO 1, during 5 years of recruitment, 88 patients treated with ustekimunab, 34 treated with vedolizumab, and 2 exposed to tofacitinib were included); however, this registry involved over 60 Spanish centres and it is a paramount study providing with data on the safety of drugs during pregnancy, as patients with this condition are excluded from clinical trials. In this regard, no sample size estimation was made, as we plan to include all patients who meet the inclusion criteria and consent their enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age diagnosed with IBD.
* Confirmed pregnancy.
* - Treatment with non-anti-TNF biologics or other advanced therapies (i.e JAK inhibitors, S1P receptor modulators and molecules approved in the forthcoming years).

Exclusion Criteria:

* Patients who do not accept to participate in the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — - Confirmed pregnancy.
Study Population: This is an observational study where pregnant women treated with non-anti-TNF agents or targeted small molecules approved for IBD treatment will be included. Although it is a multicentre, nationwide study, the number of patients to be included is expected to be relatively low (in DUMBO 1, during 5 years of recruitment, 88 patients treated with ustekimunab, 34 treated with vedolizumab, and 2 exposed to tofacitinib were included); however, this registry involved over 60 Spanish centres and it is a paramount study providing with data on the safety of drugs during pregnancy, as patients with this condition are excluded from clinical trials. In this regard, no sample size estimation was made, as we plan to include all patients who meet the inclusion criteria and consent their enrolment.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2030-05-20 (Estimated); Study Completion 2030-05-20 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of new drugs (non-anti-TNF biologics and targeted small molecules) used for IBD treatment both for pregnancy and in offspring, mainly focused on the risk of serious infections (from birth and in the first 4 years of life). | 4 years
  The measure is, number of participants with serious adverse events (all patients included should be treated with the IBD drug). And compare number of mothers with serious adverse event with differents treatments groups.

SECONDARY OUTCOMES:
To know the risk of serious adverse events (including abortions) during pregnancy and delivery associated with new drugs used for the treatment of IBD. | 4 years
To assess the developmental status of children born from IBD mothers treated with new drugs during the first 4 years of life. | 4 years
  The clinicians will complete the ASQ-3 escale. To assess children developmental status.
To compare the relative risk of serious adverse events in children born from mothers with IBD who have been exposed in utero to different new drugs to treat IBD with that of children who were not exposed to these agents. | 4 years
To compare the prevalence of malformations in children exposed to new drugs to treat IBD in utero with that of children who were not exposed to these agents. | 4 years
  To calculate the proportion of children with congenital malformations (based on the definition of the Wordld Health Organization) based on the mothers´treatment.
To evaluate the relative risk of developing neoplasm in children exposed to new drugs to treat IBD. | 4 years
  To calculate the proportion of children with neoplasm based on the mothers´ treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided